CLINICAL TRIAL: NCT07073183
Title: A Phase I Dose-Finding Study to Evaluate Safety and Tolerability of CVHNLC Plus Pembrolizumab in Patients With Squamous Non Small-Cell Lung Cancer (sqNSCLC)
Brief Title: Safety and Tolerability of CVHNLC Plus Pembrolizumab in Patients With Squamous Non Small-Cell Lung Cancer (sqNSCLC)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CV-HNLC-001; 2024-519651-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Squamous NSCLC

STUDY DESIGN:
Intervention Model Description: Phase I
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Dose escalation: CVHNLC Dose level -1 (Experimental): Dose level -1 represents a dose that may be evaluated if dose level 1 is poorly tolerated. No dose de-escalation below this level is planned for this study
  Interventions: Biological: CV09070101 mRNA vaccine (CVHNLC) 50 µg
- Dose escalation: CVHNLC Dose level 1 (Experimental)
  Interventions: Biological: CV09070101 mRNA vaccine (CVHNLC) 100 µg
- Dose escalation: CVHNLC Dose level 2 (Experimental)
  Interventions: Biological: CV09070101 mRNA vaccine (CVHNLC) 200 µg
- Dose escalation: CVHNLC Dose level 3 (Experimental)
  Interventions: Biological: CV09070101 mRNA vaccine (CVHNLC) 400 µg
- Dose expansion (Experimental): After completion of the dose-escalation part and safety data review by the DSMB, approximately 20 patients will be enrolled at the selected Recommended Dose for Expansion (RDE) to generate more data on safety, tolerability and immunogenicity.
  Interventions: Biological: CV09070101 mRNA vaccine (CVHNLC) 400 µg

INTERVENTIONS:
Biological: CV09070101 mRNA vaccine (CVHNLC) 50 µg — CVHNLC will be administered as in IM injection (4x in induction treatment period, than during main treatment period every 3 weeks) plus pembrolizumab (3-weekly)
  Arms: Dose escalation: CVHNLC Dose level -1
Biological: CV09070101 mRNA vaccine (CVHNLC) 100 µg — CVHNLC will be administered as in IM injection (4x in induction treatment period, than during main treatment period every 3 weeks) plus pembrolizumab (3-weekly)
  Arms: Dose escalation: CVHNLC Dose level 1
Biological: CV09070101 mRNA vaccine (CVHNLC) 200 µg — CVHNLC will be administered as in IM injection (4x in induction treatment period, than during main treatment period every 3 weeks) plus pembrolizumab (3-weekly)
  Arms: Dose escalation: CVHNLC Dose level 2
Biological: CV09070101 mRNA vaccine (CVHNLC) 400 µg — CVHNLC will be administered as in IM injection (4x in induction treatment period, than during main treatment period every 3 weeks) plus pembrolizumab (3-weekly)
  Arms: Dose escalation: CVHNLC Dose level 3
Biological: CV09070101 mRNA vaccine (CVHNLC) 400 µg — CVHNLC will be administered as in IM injection (4x in induction treatment period, than during main treatment period every 3 weeks) plus pembrolizumab (3-weekly) and carboplatin/paclitaxel (3-weekly)
  Arms: Dose expansion

SUMMARY:
This is an open-label, first-in-human, dose escalation study of CV09070101 mRNA (CVHNLC) in patients with metastatic Squamous Non-Small-Cell Lung Cancer (sqNSCLC).

The study will evaluate the safety and tolerability of CVHNLC plus pembrolizumab in an Dose Escalation Part and, once the safety of this combination is established, CVHNLC plus prembrolizumab and chemotherapy (carboplatin and paclitaxel) will be evaluated in an Dose Expansion Part with the recommended dose selected from the Dose Escalation Part.

DETAILED DESCRIPTION:
Dose Escalation (Metastatic 1L Maintenance sqNSCLC) The Dose Escalation Part will be comprised of 3 dose cohorts with a starting dose of 100 μg (dose level 1). Once the starting dose is established as safe, further dose levels of 200 μg and 400 μg may be explored. Depending on safety assessment guided by a Bayesian Logistic Regression Model (BLRM) design intermediate dose levels may be explored. In case the HTD is exceeded at 100 μg, a lower dose level of 50 μg may be explored.

Approximately 3 to 6 patients will be enrolled per dose level/cohort. To better understand the safety and tolerability of CVHNLC, additional patients may be enrolled in enrichment cohorts at dose levels that have previously been determined to be safe in at least 3 patients. This may be before or while proceeding with the next higher dose. An enrichment cohort may have up to 10 patients enrolled.

Each dose level will start with the staggered enrollment of 3 patients. There will be a 2-week interval between the first CVHNLC administration of the first patient and the first CVHNLC administration of the second patient. The same approach will be used between the second and third patient. If the cohort is enriched with further patients, subsequent patients may be treated concurrently once the second patient has completed the 2 weeks after the first CVHNLC administration. The enrollment is followed by a safety data review by the Safety Review Team (SRT) after all patients in each cohort have completed their 4 weeks DLT evaluation period. Non-evaluable patients (patients that discontinue/withdraw during the DLT assessment period for a reason other than DLT) may be replaced.

Safety will be continuously monitored by the Sponsor's Safety Physician, Sponsor's Medical Responsible Person (MRP) and the medical monitor with a focus on DLTs, Grade ≥ 3 AEs occurring after the DLT period, SAEs, and AESIs. After completion of the DLT evaluation period in all patients enrolled in a dose cohort, the SRT will review the safety data from the respective and all previous dose cohorts together with the Coordinating Investigator and decide about the next steps e.g.:

* Escalation of the dose to the next level.
* Enrollment of additional patients at the same or lower dose level.
* Stop or pause enrollment in the Dose Escalation Part of the trial.

At the end of the Dose Escalation Part, an independent Data Safety Monitoring Board (DSMB) will recommend a dose for the Dose Expansion Part (RDE) based on review of the complete safety data from the Dose Escalation Part and the Sponsor will decide on the RDE.

Dose Expansion Part (Metastatic 1L sqNSCLC) The optional Dose Expansion Part will include patients with histologically confirmed metastatic sqNSCLC not amenable for surgical or locoregional therapy and eligible for 1L treatment with pembrolizumab and platinum-based chemotherapy (carboplatin/paclitaxel). Patients should not have received any prior systemic treatment for metastatic disease. Previous (neo-)adjuvant treatment is only permitted if there are at least 12 months between end of such treatment and development of metastatic disease. Patients will receive CVHNLC plus 4 cycles of carboplatin and paclitaxel and pembrolizumab (3-weekly) followed by pembrolizumab maintenance therapy. Patients who discontinue prematurely from chemotherapy due to toxicity may continue on CVHNLC plus pembrolizumab. The first dose of CVHNLC will be administered one week prior to chemotherapy to avoid the immune suppressive effect from concomitant administration of steroids as premedication/supportive medication to chemotherapy treatment. Once chemotherapy is completed, CVHNLC administration will be aligned with pembrolizumab treatment to reduce patient visit burden.

The Dose Expansion Part will start with a safety lead-in, where the first 6 patients will be evaluated with focus on treatment-related AEs, SAEs, and AESIs after having completed the Day 29 visit, before continuing the enrollment. The safety data will be reviewed by the SRT and in addition by the DSMB, which will give a recommendation on dosage for treatment continuation. Patients will receive CVHNLC plus pembrolizumab for up to 12 months or until disease progression or undue toxicity. Patients not progressing after this period may continue on pembrolizumab outside of the trial according to standard of care.

ELIGIBILITY:
Inclusion Criteria:

Dose Escalation Part (Metastatic 1L Maintenance sqNSCLC)

1. Patients with histologically confirmed metastatic Stage IV (per American Joint Commission on Cancer (AJCC) Staging Manual, Eighth Edition) sqNSCLC not amenable for surgical or locoregional therapy.
2. Patients who have received pembrolizumab for 3 months but no longer than 6 months from start of pembrolizumab treatment (at least 3 cycles with a total dose of 600 mg), either as monotherapy or in combination with at least 2 cycles of chemotherapy with carboplatin and (nab-)paclitaxel as first-line treatment with no documented disease progression and who are indicated for maintenance therapy with pembrolizumab.
3. Patients able to tolerate further anti-PD-1 therapy i.e., no criteria for permanent discontinuation of pembrolizumab due to toxicity have been met during previous treatment.
4. No known targetable molecular aberration.
5. Patients having measurable disease according to RECIST 1.1.

Dose Expansion Part (Metastatic 1L sqNSCLC)

1. Patients with histologically confirmed metastatic sqNSCLC (AJCC Staging Manual, Eighth Edition) not amenable for surgical or locoregional therapy and being eligible for first-line treatment with pembrolizumab and chemotherapy with carboplatin and paclitaxel. Patients should not have received any prior systemic treatment for metastatic disease. Previous (neo-)adjuvant treatment is allowed if there are at least 12 months between end of this treatment and development of metastatic disease.

Inclusion Criteria applying to both Parts

1. Available formalin-fixed paraffin-embedded (FFPE) tumor tissue samples from non- irradiated lesions that are not older than 6 months for retrospective assessment of antigen expression and potential other biomarker analyses (in total 15 slides of at least 5 μm thickness or equivalent amount provided as a single block).
2. Recovered from all AEs related to prior therapies including anti-PD-(L)1 inhibitor treatment-related AEs to CTCAE Grade ≤ 1 or baseline (except for alopecia areata, vitiligo, chemotherapy induced polyneuropathy or endocrinopathies that are compensated by hormone replacement and Grade 2 lymphopenia).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Age ≥ 18 years on date of signing informed consent form (ICF).
5. Each patient must voluntarily sign and date an ICF approved by an Independent Ethics Committee (IEC), prior to the initiation of any, screening or trial-specific procedures.
6. Life expectancy ≥ 6 months.
7. Females who are post-menopausal (no menses for at least 12 months before the Screening Visit), or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

   Females of childbearing potential must:
   1. Have a negative serum pregnancy test (hCG) with a sensitivity of at least 25 mIU/mL within 10 to 14 days, and within 24 hours prior to starting the trial treatment a negative urine pregnancy test if serum pregnancy test not done within 24 hours prior to starting the trial treatment.
   2. Agree to ongoing pregnancy testing during the trial.
   3. Use effective contraception at least 28 days before starting trial treatment through 30 days after the last dose of trial treatment. Effective methods of birth control include:

      * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

        * oral
        * intravaginal
        * transdermal
      * Progestogen-only hormonal contraception associated with inhibition of ovulation:

        * oral
        * injectable
        * implantable
      * Intrauterine device
      * Intrauterine hormone-releasing system
      * Bilateral tubal ligation
      * Vasectomized partner + barrier method
8. Male patients, even if surgically sterilized (e.g., status post vasectomy), must:

   1. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal (coitus interruptus), spermicides only and lactational amenorrhea method are not acceptable methods of contraception.
   2. Agree to practice effective barrier contraception (condom) during the entire trial treatment period and through to 3 months after the last dose of trial treatment if their partner is of childbearing potential, even if they have had a successful vasectomy.
9. Male patients must refrain from sperm donation and female patients of childbearing potential must refrain from egg donation during the entire trial treatment period and through to 3 months after the last dose of trial treatment.
10. Able to understand the requirements of the trial and comply with the trial protocol procedures.

Exclusion Criteria:

1. Disease progression on or within 12 months after the last dose of (neo-)adjuvant anti PD-(L)1 treatment before start of first-line treatment.
2. Prior radiotherapy within 2 weeks before start of trial treatment.
3. History of other malignancies unless the patient has undergone potentially curative treatment without evidence of recurrence within the last 3 years. Exception is BCC or carcinoma in situ of any site that has been adequately treated (with the exception of systemic therapy).
4. Previous anaphylactic or severe allergic reaction to LNP-formulated drug or (mRNA) vaccine (or known allergy to any other component of CVHNLC).
5. Allergy to aminoglycoside or beta-lactam antibiotics.
6. History of previous permanent discontinuation of anti-PD-(L)1 therapy due to toxicity or any other contraindications to treatment with pembrolizumab, including severe hypersensitivity to anti-PD-1 checkpoint inhibitors, its active substance, or one of its excipients.
7. Abnormal (≥ Grade 2 NCI-CTCAE v5.0) laboratory values as follows:

   1. Hemoglobin < 10 g/dL (6.2 mmol/L).
   2. White blood cell (WBC) count decrease < 2.5 ×109/L.
   3. Absolute neutrophil count (ANC) decrease < 1.5 ×109/L.
   4. Absolute lymphocyte count (ALC) decrease < 0.5 ×109/L.
   5. Platelet count decrease < 75 ×109/L.
   6. Bilirubin > 1.5 × upper limit of normal (ULN according to the performing lab's reference range), except for patients with Gilbert's syndrome.
   7. Alanine aminotransferase (ALT) > 3 × ULN (or ≤ 5 in patients with liver metastasis).
   8. Aspartate aminotransferase (AST) > 3 × ULN. (or ≤ 5 in patients with liver metastasis).
   9. Serum creatinine increased > 1.5 × ULN or creatinine clearance < 50 mL/min.
   10. Serum Albumin < 30 g/L.
8. Received steroid treatment with doses exceeding 10 mg prednisolone or equivalent per day within 3 days prior to enrollment and/or requiring continued treatment with steroid doses above 10 mg/day prednisolone or equivalent or any other systemic immunosuppressive treatment within 28 days prior to enrollment or requiring chronic immunosuppression with such treatment. Inhalation steroids or topical steroids are allowed.
9. Active infections requiring antibiotic treatment, associated with fever > 38°C or expected to potentially result in severe disease.
10. Patients with known active hepatitis B (presence of HBsAg) or hepatitis C (presence of Hep C Ab) at screening or within 3 months prior to first trial treatment. In case of positive Hep C Ab, subjects may be enrolled in case of a negative confirmatory hepatitis C virus (HCV) RNA polymerase chain reaction (PCR) test.
11. Patients with seropositivity of human immunodeficiency virus (HIV).
12. Active autoimmune diseases (except for vitiligo or autoimmune thyroid disease that is stable under treatment), requiring treatment with steroids, disease modifying agents or immunosuppressants.
13. Brain metastases or evidence of leptomeningeal tumor spread (with exception of stable brain metastases controlled by radiotherapy or other treatment without need for steroid treatment).
14. Immunosuppression other than related to prior treatment of malignancy (i.e., platinum-based chemotherapy).
15. Previous hematopoietic stem cell or solid organ transplantation.
16. Any condition that in the judgment of the Investigator is likely to prevent compliance with trial procedures.
17. Previous immune-mediated pneumonitis, myocarditis, immune-mediated hepatitis, encephalitis or Guillain-Barré syndrome of any grade, any occurrence of a ≥ Grade 3 immune-mediated AE during previous treatment with pembrolizumab (with the exception of endocrinopathies stable under hormone replacement).
18. Patients with impaired coagulation or any bleeding disorder in whom an intramuscular injection or blood draw is contraindicated.
19. History of myocarditis or pericarditis within the last 6 months or history of myocarditis or pericarditis following mRNA COVID-19 vaccination.
20. Previous prophylactic mRNA vaccination (e.g., SARS-CoV2) or live attenuated vaccination within 30 days prior to first administration of CVHNLC treatment and other vaccines within 2 weeks prior to first administration of CVHNLC treatment.
21. Previous anticancer vaccine administrations.
22. Serious illness or condition, which according to the Investigator poses an undue risk for the patient when participating in the trial, including, but not limited to, any of the following:

    1. Clinically significant cardiovascular disease (myocardial infarction or stroke within the last 6 months, uncontrolled angina within last 3 months, diagnosed or suspected clinically significant ventricular arrhythmias, ejection fraction < 45%, cerebrovascular event within last 6 months, uncontrolled hypertension [blood pressure > 160 mmHg systolic and 100 mmHg diastolic despite] medication).
    2. New York Heart Association (NYHA) Class III to IV congestive heart failure.
    3. Symptomatic peripheral vascular disease.
    4. Severe pulmonary disease (e.g., severe chronic obstructive pulmonary disease or pulmonary fibrosis), active or history of non-infectious pneumonitis or interstitial lung disease requiring steroids.
23. Uncontrolled diabetes (repeated episodes of severe hypo- or hyperglycemia requiring hospitalization).
24. Severe mental retardation/impairment, psychiatric conditions or substance abuse resulting in inability to understand informed consent or affecting patient's cooperation in the trial.
25. Pregnant or breastfeeding patients.
26. Concurrent or prior (within 30 days or at least 5 half-lives of investigational product, whatever is longer prior to trial enrollment) participation in another investigational clinical trial studying an investigational product or treatment regimen.
27. Patients with any contraindications to the SOC/AxMP as detailed in the approved product label or SmPC/USPI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events (TRAEs) | 1 year
Incidence of treatment-emergent adverse events (TEAEs) | 1 year
Incidence of serious adverse events (SAEs) | 1 year
Incidence of adverse events of special interest (AESIs) | 1 year
Incidence of immune-related adverse events (irAEs) | 1 year
Incidence of injection site reactions (ISRs) | 1 year
Incidence of medical attended adverse events (MAEs) treatment-emergent adverse events leading to treatment discontinuation | 1 year
Incidence of clinically significant laboratory abnormalities per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.5.0. | 1 year
Number of patients with dose-limiting toxicities (DLTs) evaluated during the first 4 weeks of treatment (Dose Escalation Part only) | 1 year

SECONDARY OUTCOMES:
Objective response rate based on best overall response assessed by the Investigator using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1). Response is defined as patients achieving either a complete response (CR) or partial respo | 1 year
Progression-free survival (PFS) based on RECIST 1.1. Response is defined as time from first trial treatment to time of disease progression or death due to disease progression | 1 year
Duration of response per RECIST 1.1, measured from the time of first documentation of response until first documentation of disease progression. | 1 year
Disease control rate (DCR) at 3, 6, 9 and 12 months based on RECIST 1.1. Disease control is defined as stable disease (SD), partial response (PR) or complete response (CR). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Information, Study Director — CureVac SE
Locations (13):
- United States (2):
  - Virginia Cancer Center, Fairfax, Virginia
  - Virginia Commonwealth University, Massey Comprehensive Cancer Center, McGlothlin Medical Education Center, Richmond, Virginia
- France (6):
  - AP-HM - Hôpital Nord, Marseille
  - Institut Curie - Hôpital de Paris, Paris
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - Institut de Cancerologie de l'Ouest - Hôpital Saint Herblain - PPDS, Saint-Herblain
  - Institut Claudius Regaud - PPDS, Toulouse
  - Gustave Roussy, Villejuif
- Spain (5):
  - Hospital Quironsalud Barcelona -NEXT Oncology, Barcelona, Spain
  - Hospital Universitari Vall d´Hebron -Instituto de Investigacion Oncologica Vall dHebron (VHIO), Barcelona, Spain
  - Hospital Universitario Fundacion Jimenez Diaz - START MADRID, Madrid, Spain
  - Hospital Universitario HM Sanchinarro - CIOCC - START MADRID, Madrid, Spain
  - Hospital Regional Universitario Virgen de la Victoria, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No